CLINICAL TRIAL: NCT01804582
Title: The Family VOICE Study (Value, Information, Community Support, and Experience): A Randomized Trial of Family Navigator Services Versus Usual Care for Care of Young Children Treated With Antipsychotic Medication
Brief Title: The Family VOICE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Gloria Reeves, M.D. , Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00054913; 1300476 (Other: Patient Centered Outcome Research Institute (PCORI))
Record Dates: First submitted 2013-02-27; First posted 2013-03-05 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Autism; Aggression; Bipolar Disorder; Psychotic Disorders
Keywords: Family navigator; Patient Centered Outcomes; Pediatric Antipsychotic treatment
MeSH Terms: conditions — Autistic Disorder; Aggression; Bipolar Disorder; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Navigator Consultation (Experimental): This group of parents will be contacted by a Family Navigator to assist them in accessing psychosocial resources based on their child and family needs. Components of this intervention are the following:
  (1)family engagement; (2) inquiry about psychosocial resource needs related to schools, outpatient child treatment, support programs, or mental health resources for other household family members; (3) discuss potential benefits/challenges of options and parent preferences/priorities for care; (4) assessment on perceived barriers to seeking resources; (5) collaborative problem solving to address barriers; (6) discuss options for follow up plan.
  Interventions: Other: Family Navigator consultation
- Usual Care (No Intervention): No specific study intervention is provided to this group of parents. This control group will received the usual care that they have been receiving from their child's providers.

INTERVENTIONS:
Other: Family Navigator consultation — Telephone contact from the trained family navigator to the parent participant several times over the 90 day study time period. Components of the service include the following:
  (1)family engagement; (2) inquiry about psychosocial resource needs related to schools, outpatient child treatment, support programs, or mental health resources for other household family members; (3) discuss potential benefits/challenges of options and parent preferences/priorities for care; (4) assessment on perceived barriers to seeking resources; (5) collaborative problem solving to address barriers; (6) discuss options for follow up plan.
  Other Names: Patient navigator services
  Arms: Family Navigator Consultation

SUMMARY:
Family centered mental health treatment with children values and supports the role of parents in their child's recovery. However, medications are often the primary focus in community treatment, even in preschool age youth, with increasing use of antipsychotic medication for serious mood and behavior problems. Although medication may be necessary to address safety issues (such as severe aggression) it can cause serious side effects, such as obesity, and medication only does not follow recommended care for these types of problems. Psychosocial treatments are highly recommended (e.g. Programs that coach empower parents to manage their child's difficult behaviors) as part of comprehensive child treatment. Parent involvement in psychosocial treatment has clear benefits for their child's mental health, and unlike medication, the effects can last long after treatment is completed. However, problems related to access (e.g. long waiting lists) and use (e.g. parent mistrust mental health services) of services are common. Maryland, like other states, has developed a system to improve medication safety by reviewing health information about the child to determine if the treatment is appropriate. This reduces unnecessary medication treatment and ensures children have adequate health screening before starting any treatment. Those approved for medication have moderate-severe mental health problems, which supports their need for comprehensive (medication and psychosocial) treatment, instead of medication only. In this study, investigators partner with parents/family advocates, child-serving agencies, and health providers to develop a Family Navigator (FN) Service to link with this medication program. A FN is an individual who has cared for their own child with mental illness. The FN supports parents, provide information on psychosocial treatment options, and address barriers to using services. The goals of this program are to improve use of psychosocial services, and to improve parent empowerment, support, and satisfaction with their child's mental health treatment. The investigators also expect that the FN Service will improve the child's overall mental health and reduce the likelihood of a medication dose increase or another medication added during the initial treatment period. The FN Service is provided for parents of public insured children ages 3-15 years newly approved for antipsychotic medication treatment. The FN Services will be provided by phone, which supports families in both rural and urban settings. The investigators' long term goal is to develop a FN program that strongly supports Family-centered treatment of children and can be used to help families in other underserved areas beyond Maryland.

DETAILED DESCRIPTION:
Background: Emerging data on serious antipsychotic medication side effects (e.g. new onset diabetes)has heightened concerns about sharp increases in "off label" pediatric antipsychotic treatment of mood/behavioral disorders, and led to increased scrutiny of pediatric mental health treatment. Several states are developing antipsychotic medication pre-authorization programs to reduce inappropriate or unsafe prescribing. This Healthcare system change, however, fails to address a critical underlying problem that parents are not effectively engaged to utilize non-medication treatments and serve an active role in their child's mental health recovery. Psychosocial treatments (e.g. parenting skills training to manage aggressive behaviors) are evidence-based interventions that are poorly utilized in community care. The Maryland Medicaid program developed a pediatric Antipsychotic Pre-Authorization Program that requires providers to make at least one psychosocial treatment referral in order to obtain medication approval. This program was shaped by strong input from parents, health experts, and child serving agency administrators to promote psychosocial treatment referral, but it does not provide any Family-centered services to improve treatment utilization. Objectives: We propose to link the Antipsychotic Pre-Authorization Program with a Family Navigator Service. The investigators will examine if Navigator Services improve parent empowerment, support, and satisfaction with child services. The investigators will also assess if Navigator Services are associated with improved psychosocial service utilization, improved child functioning, and lower likelihood of medication increases (higher dose or addition of another medication). The investigators' long term objective is to develop a Family Navigator model that is highly portable, amenable for use in underserved areas, addresses the needs of low income families with young children, and promotes evidence-based mental health care. Methods: The investigators will conduct a randomized trial of a telephone Family Navigator Service versus usual care for 240 Medicaid insured youth 10 years old who are approved for antipsychotic medication treatment. The Family Navigator is a parent who has experienced their own child's mental illness. Navigators will provide support, information on psychosocial treatment options, and options to address barriers to care. The investigators will assess family-centered outcomes at baseline and 90 days (medication re-authorization). The investigators will use generalized linear mixed effects models with the appropriate link functions to assess whether there is a significant difference in improvement from baseline to the post-treatment assessment on the outcome variables between the Family Navigator condition and treatment as usual condition. A significant interaction between time and study condition would support the hypothesis that a Family Navigator will improve parent and child outcomes.

ELIGIBILITY:
Inclusion Criteria:

Child 2 to 15 years old who has been approved by the Maryland Medicaid program for treatment with an antipsychotic medication.

Exclusion Criteria:

Department of social services custody

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria M Reeves, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, School of Medicine, Department of Psychiatry, Division of Child and Adolescent Psychiatry, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olin SS, Hoagwood KE, Rodriguez J, Radigan M, Burton G, Cavaleri M, Jensen PS. Impact of Empowerment Training on the Professional Work of Family Peer Advocates. Child Youth Serv Rev. 2010 Oct 1;32(10):1426-1429. doi: 10.1016/j.childyouth.2010.06.012. PMID 21076659

RESULTS

PARTICIPANT FLOW:
Groups:
- Family Navigator Consultation: Family Navigator consultation: Telephone contact from the trained family navigator to the parent participant several times over the 90 day study time period. Components of the service include the following:
  (1)family engagement; (2) inquiry about psychosocial resource needs related to schools, outpatient child treatment, support programs, (3) discuss potential benefits/challenges of options and parent preferences/priorities for care;(4) assessment on perceived barriers to seeking resources; (5) collaborative problem solving to address barriers; (6) discuss options for follow up plan.
Period: Overall Study
Arm/Group | Family Navigator Consultation | Usual Care
Started | 177 | 173
Completed | 128 | 117
Not Completed | 49 | 56
Not completed — Lost to Follow-up | 47 | 56
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Population: Two participants were removed from the study after they were found to be ineligible due to not being the parent/legal guardian. This decreased our Family Navigator Group from 177 to 175 participants. The Usual Care group remained the same at 173 for a total sample size of N = 348.
Groups:
- Family Navigator Consultation: Family Navigator consultation: Telephone contact from the trained family navigator to the parent participant several times over the 90 day study time period. Components of the service include the following:
  (1)family engagement; (2) inquiry about psychosocial resource needs related to schools, outpatient child treatment, support programs, (3) discuss potential benefits/challenges of options and parent preferences/priorities for care; (4) assessment on perceived barriers to seeking resources; (5) collaborative problem solving to address barriers; (6) discuss options for follow up plan.
- Total: Total of all reporting groups
Arm/Group | Family Navigator Consultation | Usual Care | Total
Number analyzed (Participants) | 175 | 173 | 348
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 170 | 168 | 338
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.09 (10.06) | 38.47 (10.00) | 39.28 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 158 | 325
  Male | 8 | 15 | 23
Region of Enrollment [Number; unit: participants]
  United States | 175 | 173 | 348

OUTCOME MEASURES:

1. Primary Outcome: Family Empowerment Scale
Description: This 34-item, Likert scale with scores ranging from 1 (never) to 5 (very often) which measures parent empowerment related to caring for their child with special needs. Higher scores indicate a greater sense of parental empowerment in caring for their child, interacting with the services system and contributing to the community. The sub scales have demonstrated good reliability and validity, and provide comprehensive information about empowerment, including attitudes, knowledge, and behaviors. A composite score was calculated for each participant with the range 1-5 (1 never to 5 very often)based on the average of their item scores with higher scores indicating better outcomes.
Time Frame: Change from baseline to 90 days
Population: An intent to treat analysis was conducted with a linear mixed model which included data from all participants collected at baseline and 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family Navigator Consultation | Usual Care
Number analyzed (Participants) | 175 | 173
units on a scale
  baseline outcome | 3.75 (.52) | 3.86 (.51)
  3 month outcome | 3.81 (.55) | 4.02 (.51)
Statistical Analysis 1: Comparison: Family Navigator Consultation vs Usual Care; An intent to treat analysis was conducted using a linear mixed model to determine if there was any significant difference in change from baseline to 3 months based on time and condition. Data for all participants was included at baseline and 3 months; Test type: Superiority or Other; p = .15, Mixed Models Analysis

2. Primary Outcome: Duke-UNC (University of North Carolina) Functional Social Support Questionnaire
Description: This 14 item questionnaire assesses confidant ("e.g. "I get chances to talk to someone I trust about family problems."), affective ("People care what happens to me."), and instrumental ("I can get help when I need transportation support."). In a validation sample, the measure was found to have good internal consistency and it correlated with related domains of psychosocial functioning in expected directions. This measure has been widely used to assess social support among both identified medical and mental health patients as well as their family members. A composite score was calculated for each participant with the range 1-5 (1 As much as I would like to 5 Much less than I would like) based on the average of their item scores. The range of scores is from 1-5 with lower scores indicating better functional social support. Subscales were not analyzed.
Time Frame: Change from Baseline to 90 days
Population: An intent to treat analysis was conducted with a linear mixed model on all outcome data collected at baseline and 3 months to determine significance of change.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Family Navigator Consultation: This group of parents will be contacted by a Family Navigator to assist them in accessing psychosocial resources based on their child and family needs. Components of this intervention are the following:
  (1)family engagement; (2) inquiry about psychosocial resource needs related to schools, outpatient child treatment, support programs, or mental health resources for other household family members; (3) discuss potential benefits/challenges of options and parent preferences/priorities for care; (4) assessment on perceived barriers to seeking resources; (5) collaborative problem solving to address barriers; (6) discuss options for follow up plan.
  Family Navigator consultation: Telephone contact from the trained family navigator to the parent participant several times over the 90 day study time period. Components of the service include the following:
  (1)family engagement; (2) inquiry about psychosocial resource needs related to schools, outpatient child treatment, support programs,
Arm/Group | Family Navigator Consultation | Usual Care
Number analyzed (Participants) | 175 | 173
units on a scale
  Baseline Outcome | 2.58 (1.10) | 2.46 (1.07)
  3 month Outcome | 2.48 (1.10) | 2.45 (1.06)
Statistical Analysis 1: Comparison: Family Navigator Consultation vs Usual Care; Test type: Superiority or Other; p = .53, Mixed Models Analysis; Mean Difference (Final Values) = .07 — Cohen's d was calculated to measure the estimation parameter

3. Primary Outcome: Youth Services Survey for Families
Description: This 26-item questionnaire specifically targets parents' satisfaction with children's mental health services. The measure assesses five domains of parent satisfaction: cultural sensitivity, access, treatment participation, appropriateness, and outcome. This measure has been adopted by several State mental health systems to evaluate parent satisfaction with child services. A composite score was calculated for each participant with the range 1-5 (1 Strongly Disagree to 5 Strongly Agree) based on the average of their item scores. Range of scores is from 1-5 with higher scores indicating better functional social support. Subscales were not analyzed.
Time Frame: Change from Baseline to 90 days
Population: An intent to treat analysis was conducted with a linear mixed model on all data collected at baseline and 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family Navigator Consultation | Usual Care
Number analyzed (Participants) | 175 | 173
units on a scale
  Baseline Outcome | 3.75 (.64) | 3.90 (.63)
  3 month Outcome | 3.81 (.61) | 3.95 (.60)
Statistical Analysis 1: Comparison: Family Navigator Consultation vs Usual Care; Test type: Superiority or Other; p = .80, Mixed Models Analysis; Mean Difference (Final Values) = .03

4. Secondary Outcome: Child Behavior Checklist - Brief Problem Monitor
Description: We will use the preschool (ages 1 ½-5) and school age (6-12) versions of this measure, which asks parents to rate items about behavioral and emotional problems on a 0-2 scale. Both versions provide a Total Problem Score. These measures have been widely used in pediatric mental health research. The Brief Problem Monitor provides T scores for the total problem score and it ranges from 0-80, with higher T scores indicating more mental health difficulties. Subscales of this measure were not analyzed.
Time Frame: Change from Baseline to 90 days
Population: An intent to treat analysis was conducted with a linear mixed model on all data collected at baseline and 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family Navigator Consultation | Usual Care
Number analyzed (Participants) | 175 | 173
units on a scale
  Baseline Outcome | 69.51 (5.69) | 69.19 (5.62)
  3 month Outcome | 67.63 (6.03) | 66.73 (6.83)
Statistical Analysis 1: Comparison: Family Navigator Consultation vs Usual Care; Test type: Superiority or Other; p = .33, Mixed Models Analysis

5. Secondary Outcome: Psychosocial Service Utilization
Description: We will utilize total Medicaid claims data for any psychosocial services claims (e.g. individual, family, or group psychotherapy; parenting groups) to collect information on services used in the 90 days prior to the baseline and over the 90 days of participant enrollment in the study. Participants were considered to have received psychosocial claims (dichotomous Yes/No) if they received any individual, family, or group psychotherapy in the 90 days prior and during the study period. Higher numbers indicate more participants received at least 1 psychosocial service claim.
Time Frame: Change from Baseline to 90 days
Population: The same participants 175 FN and 173 TAU participants were analyzed for psychosocial claims during the 90 day period prior to enrollment and then 90 days during enrollment. The count of participants represents the number of subjects (from the 175 FN and 173 TAU) that had at least 1 claim during each specified time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Family Navigator Consultation | Usual Care
Number analyzed (Participants) | 175 | 173
Participants
  PS claim 90 days prior to enrollment with services | 120 | 108
  90 days during enrollment | 112 | 108
  No PS claim 90 day prior to enrollment | 35 | 65
  No PS claim 90 days during enrollment | 63 | 65
Statistical Analysis 1: Comparison: Family Navigator Consultation vs Usual Care; Test type: Superiority or Other; p = .21, Wald Chi-Squared

6. Secondary Outcome: Medication Regimen
Description: We will utilize Medicaid pharmacy prescription data collect information at baseline and 90 days on the name and dose of all psychiatric medications prescribed at those time points. Participants were designated increase or no increase in their dosage of antipsychotic medication (i.e., dichotomous Yes/No) over the 90 day intervention period.
Time Frame: Change from Baseline to 90 days
Population: The total n=229 included those on medication at 90 days (119 never filled the prescription or changed to a different med).
Measure: Count of Participants; unit: Participants
Arm/Group | Family Navigator Consultation | Usual Care
Number analyzed (Participants) | 110 | 119
Participants
  Dose increase over 90 days | 26 | 49
  No dose increase over 90 days | 84 | 70
Statistical Analysis 1: Comparison: Family Navigator Consultation vs Usual Care; The total n=229 included those on medication at 90 days (119 never filled the prescription or changed to a different med); Test type: Superiority or Other; p = .005, Chi-squared; Chi Squared (1, N = 229) = 7.99; Phi = .19

ADVERSE EVENTS:
Time Frame: Safety monitoring for adverse events was conducted throughout the study for each participant at baseline, each family navigator contact and 3 months. Over the course of the study 3 cases of suspected abuse was reported to the Department of Social Services Child Protective Services.
Groups:
- Family Navigator Consultation: Family Navigator consultation: Telephone contact from the trained family navigator to the parent participant several times over the 90 day study time period. Components of the service include the following: (1)family engagement; (2) inquiry about psychosocial resource needs related to schools, outpatient child treatment, support programs, or mental health resources for other household family members; (3) discuss potential benefits/challenges of options and parent preferences/priorities for care; (4) assessment on perceived barriers to seeking resources; (5)collaborative problem solving to address barriers; (6) discuss options for follow up plan.
Arm/Group | Family Navigator Consultation | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/177 | 0/173
Other Adverse Events (participants affected / at risk) | 3/177 | 0/173
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Family Navigator Consultation (N=177) | Usual Care (N=173)
Suspected Child Abuse/Neglect (Psychiatric disorders) | 3 (3) | 0 (0) — The study team is mandated by state and federal law to report any suspicion of child abuse/neglect to the Department of Social Services in the jurisdiction in which the event occurred.

LIMITATIONS AND CAVEATS:
The Family Navigator had telephone-only contact with the parent and there was not required schedule of visits. The "dosing" of the intervention may not have been sufficiently powered to impact empowerment as measured by the FES given our sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No